CLINICAL TRIAL: NCT02558270
Title: Acute Effects of Sodium GlucOse Co-Transporter 2 (SGLT2) Inhibition on Hepatic Glucose and Energy Metabolism
Brief Title: Effects of SGLT-2 Inhibition on Hepatic Glucose and Energy Metabolism
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Michael Krebs, Prof. MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GOETHE_V2
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes; Metabolically Healthy Controls
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- patients dapa (Active Comparator): Patients will be administered Dapagliflozin 10mg
  Interventions: Drug: Dapagliflozin
- patients placebo (Placebo Comparator): Patients will be administered a placebo
  Interventions: Drug: Placebo
- controls dapa (Active Comparator): controls will be administered Dapagliflozin 10mg
  Interventions: Drug: Dapagliflozin
- controls placebo (Placebo Comparator): controls will be administered a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin
  Arms: controls dapa; patients dapa
Drug: Placebo
  Arms: controls placebo; patients placebo

SUMMARY:
Inhibition of SGLT2 by specific inhibitors has been shown to reduce the renal threshold for glucose excretion in patients with type 2 diabetes mellitus (T2DM) and control subjects leading to significant renal glucose loss even in the presence of normal glucose concentrations. SGLT2 inhibition with canagliflozin induces a 24h urinary glucose loss of around 70g in healthy subjects.

Recent studies indicate that under fasting and postprandial conditions administration of SGLT-2 inhibitors leads to increase in endogenous (hepatic) glucose production (EGP) potentially counteracting the glucose lowering potency of these drugs. Dapagliflozin has been shown to acutely increase endogenous glucose production (EGP) and plasma glucagon concentrations under postabsorptive conditions within 2 hours after drug ingestion in patients with (T2DM). Glucagon binds to receptors in the liver and activates hepatic gluconeogenesis (GNG) and glycogenolysis, likely contributing to the observed increase in EGP.

So far the likely interrelation between acute changes in hepatic glucose metabolism and energy turnover contributing to increased hepatic glucose production induced by SGLT2 inhibition has not been studied. It is known that out of the 80% of oxygen consumption coupled to ATP synthesis, 7- 10% is used by GNG. However, so far the effects of dapagliflozin on acute changes in gluconeogenesis (GNG) and ATP turnover in hepatic tissue and on the time course of hormones involved in hypoglycaemia counter regulation have not been studied.

ELIGIBILITY:
Inclusion criteria for diabetic patients:

* Type 2 diabetes
* BMI 23 - 35 kg/m2
* Age between 18 - 75 years
* HbA1c < 7.5% while on dietary treatment only or treatment!with!up!to!two!oral!antidiabetic! agents!including!metformin,!alphaAglucosidase!inhibitor,!sulfonyl!urea!or!DPPAIV!inhibitor.
* Must have given written informed consent and be able to comply with all study requirements
* Males or females. Aged 18 to 75 years, inclusive, at the time of informed consent
* Females: Non-pregnant and non-lactating; surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved), abstinent, or if engaged in sexual relations of child-bearing potential, subject is using an acceptable contraceptive method.
* Body Mass Index (BMI) 23 - 35 kg/m2
* Agree to maintain current diet and exercise regimen. Agree to abstain from alcoholic beverages for at least 48 hours prior to clinic visits and not increase alcohol consumption during the study

Exclusion criteria for diabetic patients:

* smoking
* pregnancy
* treatment with more than 2 oral antidiabetic agents or treatment with insulin / SGLT2 inhibitor
* regular medication
* tendency towards claustrophobia
* metal devices or other magnetic material in or on the subjects body which will be hazardous for NMR investigation [heart pacemaker, brain (aneurysm) clip, nerve stimulators, electrodes, ear implants, post coronary by-pass graft (epicardial pace wires), penile implants, colored contact lenses, patch to deliver medications through the skin, coiled spring intrauterine device, vascular filter for blood clots, orthodontic braces, shunt-spinal or ventricular, any metal implants (rods, joints, plates, pins, screws, nails, or clips), embolization coil, or any metal fragments or shrapnel in the body].
* Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN, Total bilirubin >2.0 mg/dL (34.2 μmol/L), positive serologic evidence of current infectious liver disease including Hepatitis B viral antibody IGM, Hepatitis B surface antigen and Hepatitis C virus antibody
* Creatinine Clearance: <60 mL/min (calculated by Cockcroft-Gault formula) or a measured serum creatinine value of >1.5 mg/dL (133 μmol/L) for male patients and >1.4 mg/dL (124 μmol/L) for female patients, History of unstable or rapidly progressing renal disease
* History of diabetic ketoacidosis (DKA) requiring medical intervention (eg, emergency room visit and/or hospitalization) within 1 month prior to the Screening visit.
* Volume depleted patients.
* Recent Cardiovascular Events in a patient:

  * Acute Coronary Syndrome (ACS) within 2 months prior to enrolment
  * Hospitalization for unstable angina or acute myocardial infarction within 2 months prior to enrolment
  * Acute Stroke or TIA within two months prior to enrolment
  * Less than two months post coronary artery revascularization
* Congestive heart failure defined as New York Heart Association (NYHA) class IV, unstable or acute congestive heart failure.
* Treatment with insulin, thiazolidinedione (e.g., pioglitazone), GLP-1 agonist, SGLT2 and other drugs that may affect plasma glucose level (including systemic glucocorticoids) within 3 months prior to screening

Exclusion criteria for healthy controls:

* Clinically!significant!abnormalities!in!medical!history!or!physical!examination + smoking
* regular medication
* pregnancy, breast feeding
* tendency towards claustrophobia
* metal devices or other magnetic material in or on the subjects body which will be hazardous for NMR investigation [heart pacemaker, brain (aneurysm) clip, nerve stimulators, electrodes, ear implants, post coronary by-pass graft (epicardial pace wires), penile implants, colored contact lenses, patch to deliver medications through the skin, coiled spring intrauterine device, vascular filter for blood clots, orthodontic braces, shunt-spinal or ventricular, any metal implants (rods, joints, plates, pins, screws, nails, or clips), embolization coil, or any metal fragments or shrapnel in the body].
* Hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN, Total bilirubin >2.0 mg/dL (34.2 μmol/L), positive serologic evidence of current infectious liver disease including Hepatitis B viral antibody IGM, Hepatitis B surface antigen and Hepatitis C virus antibody
* Creatinine Clearance: <60 mL/min (calculated by Cockcroft-Gault formula) or a measured serum creatinine value of >1.5 mg/dL (133 μmol/L) for male patients and >1.4 mg/dL (124 μmol/L) for female patients, History of unstable or rapidly progressing renal disease
* Volume depleted patients. Patients at risk for volume depletion due to co-existing conditions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change in endogenous glucose production | 420 minutes

SECONDARY OUTCOMES:
Change in hepatic gluconeogenesis | 420 minutes
Change in hepatic lipid content | 420 minutes
Change in hepatic glycogen content | 420 minutes
Changes in hepatic ATP concentrations | 420 minutes
Changes in hormones involved in hypoglycemia counter regulation | 420 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Of Vienna, Department of Internal Medicine III, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Wolf P, Fellinger P, Pfleger L, Beiglbock H, Krumpolec P, Barbieri C, Gastaldelli A, Harreiter J, Metz M, Scherer T, Zeyda M, Baumgartner-Parzer S, Marculescu R, Trattnig S, Kautzky-Willer A, Krssak M, Krebs M. Gluconeogenesis, But Not Glycogenolysis, Contributes to the Increase in Endogenous Glucose Production by SGLT-2 Inhibition. Diabetes Care. 2021 Feb;44(2):541-548. doi: 10.2337/dc20-1983. Epub 2020 Dec 14. PMID 33318126